CLINICAL TRIAL: NCT02092740
Title: Retrospective Analysis of Testicular Cancer Patients With Histopathological Analysis or Urological Treatment at the University Magdeburg 1960-2012.
Brief Title: REtrospective Study of TESTIcular CAncer Patients at the University Magdeburg
Acronym: RETESTICAPUM
Status: Completed | Type: Observational
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Johann J. Wendler, MD, Dr. med. Johann Jakob Wendler, University of Magdeburg
Other Study IDs: DE-UKMD-URO-0023
Record Dates: First submitted 2014-03-14; First posted 2014-03-20 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Testicular Cancer
Keywords: Testicular cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Seminoma: Seminoma
- Non-Seminoma: Non-Seminoma

SUMMARY:
Retrospective analysis of treatment outcome and side effects of testicular cancer patients that had been diagnosed at the University Magdeburg from 1960 until 2012.

DETAILED DESCRIPTION:
Creating an ACCESS Windows form based Data Registry for testicular cancer patients.

Relevant data for testicular cancer patients based on EAU-guidelines 2013 and EORTC/RTOG, Lent-SOMA, CTC. All testicular cancer patients who had been histopathologically diagnosed al the Institute of Pathology at the University Magdeburg. About 2000 patients from 1960 until 2012. Postgraduate students collecting data requesting hospital documents, cancer registry of Sachsen-Anhalt, family practitioners and urologists as well as patients. Statistically Analysis with ACCESS and IBM SPSS statistics.

ELIGIBILITY:
Inclusion Criteria:

* testicular cancer histopathologically diagnosed at the University Magdeburg Germany

Exclusion Criteria:

* none.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Testicular cancer histopathologically diagnosed at the University Magdeburg 1960-2012
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 52 years.
  Overall survival (OS).

SECONDARY OUTCOMES:
Disease-specific survival. | Up to 52 years.
  Disease-specific survival of testicular cancer.
Chronic side effects of testicular-cancer-specific radiation therapies. | Up to 52 years.
  All Therapy Associated side effects of radiation therapy using EORTC (European Organisation for Research and Treatment of Cancer) /RTOG- (Radiation Therapy Oncology Group) - RTOG/EORTC Late Radiation Morbidity Scoring Schema), LENT-SOMA-(Late Effects of Normal Tissues)-, CTCAE-(Common Terminology Criteria for Adverse Events V4)-Scores. See
Chronic side effects of testicular-cancer-specific chemotherapies. | Up to 52 years.
  All Therapy Associated side effects of chemotherapy using CTCAE-(Common Terminology Criteria for Adverse Events V4)-Score.
Chronic side effects of testicular-cancer-specific surgical therapies. | Up to 52 years.
  All Therapy Associated side effects of surgical therapy using CTCAE-(Common Terminology Criteria for Adverse Events V4)-Score.
Secondary Malignoma | Up to 52 years.
  Assessment of Development of Secondary malignoma after diagnosis of testicular cancer; Secondary malignoma other than testicular cancer and metachronous Primary testicular cancer
Progressive-free survival (PFS). | Up to 52 years.
  Progressive-free survival (PFS).
Relapse-free survival (RLS). | Up to 52 years.
  Relapse-free survival (RLS).
Quality of Life (QoL). | Current situation.
  Assessment of the current QoL using ECOG and EORTC-QLQ-C30-V3D.
Cause of death. | Up to 52 years.
  Cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Johann J Wendler, Dr. Med., Principal Investigator — Department of Urology University Magdeburg Germany
Locations (1):
- Urology University Magdeburg, Magdeburg, Saxony-Anhalt, Germany